CLINICAL TRIAL: NCT01273194
Title: Evaluating Supportive Care for Children With Cancer: A Multi-Institutional Survey Study of Pediatric Oncology Patients and Parents
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 110063; 11-CC-0063
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2015-09-08

CONDITIONS: Pediatric Cancer
Keywords: Palliative Care; Survey; Quality of Life; Attitudes; Pediatric Cancer
MeSH Terms: conditions — Neoplasms; Behavior

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

- Palliative care, also known as comfort care, is intended to keep a patient comfortable by focusing on pain and symptom management to improve quality of life. Although palliative care has been demonstrated to be beneficial, it is underutilized in children who have been diagnosed with cancer, because current trends favor palliative care primarily at the end of life and in only a small number of patients. Children with cancer likely would benefit from the incorporation of palliative care from the time of diagnosis, but both doctors and families are often reluctant to include it for a variety of reasons. Researchers are interested in understanding these reasons to determine better ways to include palliative care as part of cancer treatment methods in children with cancer.

Objectives:

- To collect information on pediatric oncology patients and their parents attitudes towards palliative care, along with cancer treatment, from the time of diagnosis.

Eligibility:

* Children and adolescents between 10 and 17 years of age who have been diagnosed with cancer in the past year.
* Parents of eligible children.

Design:

* Participants will complete a 30-minute survey about experiences with pain, symptom management, and focus on quality of life in the first month following cancer diagnosis. Child participants will be asked about their views on the importance of quality of life in the beginning of their illness, as well as their attitudes toward symptom-oriented care. Parent participants will be asked questions about their child s illness, which includes understanding, discussion, and impact of illness.
* Treatment will not be provided as part of this protocol.

DETAILED DESCRIPTION:
Background:

* Palliative care, while demonstrated to be beneficial, is underutilized in pediatric oncology.
* The current model in the U.S. favors palliative care involvement primarily at the end of life and only in a fraction of patients.
* Children with cancer likely would benefit from the incorporation of palliative care from the time of diagnosis.
* Obstacles to the incorporation of palliative care from the time of diagnosis include the possibility that the current model provides sufficient care in these areas and the possibility that families may be averse to early palliative care involvement on the grounds that it would be intrusive, detract from their goal of cure, and/or lead to a loss of hope.
* To gather data relevant to evaluating these potential obstacles, we plan to interview pediatric oncology patients and their parents to determine their views regarding provision of palliative care, along with cancer therapy, from the time of diagnosis.

Objectives:

* Primary

  * To assess parent and patient attitudes toward the integration of palliative care in pediatric oncology patients from the time of diagnosis.
  * To develop a survey instrument that can reliably assess the views of pediatric oncology patients and their parents with regard to patients symptom burden and management at the beginning of cancer therapy as well as attitudes toward early integration of palliative care with oncology care.
* Secondary/Specific Objectives

  * To assess the degree and effect of negative symptoms in children with cancer in the beginning of cancer therapy as well as the extent to which pediatric patients symptoms and suffering at this time are being adequately managed.
  * To assess the emphasis that families place on quality of life in symptom management and treatment decision making as well as the satisfaction with the degree of attention given to quality of life by the medical team.
  * To assess patient and parent attitudes toward palliative care in general and receptivity toward pediatric palliative care team involvement from the time of diagnosis.
  * To assess understanding of prognosis and its relationship to parent and patient attitudes toward the integration of palliative care in pediatric oncology care from the time of diagnosis.
  * To assess concordance between parents and patients in their attitudes toward the integration of palliative care in pediatric oncology patients from the time of diagnosis.

Eligibility:

-Patients eligible for inclusion will be children diagnosed with an oncologic disease at least 1 month and no greater than 1 year prior with age at diagnosis of 10 to 17 years. Both patient and parent must agree to participate to be eligible for inclusion.

Design:

* Surveys will be administered to consenting patient/parent pairs with the parent completing a written survey while the patient is surveyed in the absence of the participating parent.
* Total enrollment will be a minimum of 70 subject pairs and a maximum of 110 subject pairs with a target goal of 100 subject pairs enrolled over a 6 month period.

Data collected from responses to the surveys will be analyzed at the conclusion of the survey period to assess for individual content as well as concordance between the patients and their parents.

ELIGIBILITY:
* INCLUSION CRITERIA:

Pediatric Oncology Patients:

* Current patients receiving clinical care for cancer at one of the participating sites.
* At least 1 month and no more than 1 year after initial diagnosis.
* Physically and cognitively able to participate in a 30 minute interview as determined by the primary medical providers.
* Ability to understand and speak English.
* Age 10-17 at the time of first diagnosis.
* Agreement of both parent and child to participate.

Parents:

* A parent of an eligible child
* Physically and cognitively able to complete a 30 minute self-administered survey.
* Ability to read, understand and speak English.
* Agreement of both parent and child to participate.

EXCLUSION CRITERIA:

* Inability to speak English.
* Inability to understand spoken English.
* Parent s inability to read written English.
* Lack of agreement of both parent and child to participate.

Ages: 10 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-12-20; Study Completion 2015-09-08

CONTACTS AND LOCATIONS:
Overall Officials: David Wendler, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Harris MB. Palliative care in children with cancer: which child and when? J Natl Cancer Inst Monogr. 2004;(32):144-9. doi: 10.1093/jncimonographs/lgh007. PMID 15263058
- [Background] Gatta G, Capocaccia R, Coleman MP, Ries LA, Berrino F. Childhood cancer survival in Europe and the United States. Cancer. 2002 Oct 15;95(8):1767-72. doi: 10.1002/cncr.10833. PMID 12365026
- [Background] Wolfe J, Grier HE, Klar N, Levin SB, Ellenbogen JM, Salem-Schatz S, Emanuel EJ, Weeks JC. Symptoms and suffering at the end of life in children with cancer. N Engl J Med. 2000 Feb 3;342(5):326-33. doi: 10.1056/NEJM200002033420506. PMID 10655532